CLINICAL TRIAL: NCT04643990
Title: Clinical Analysis of LDT Combined With TDF to Improve EGFR Decreasing in Patients With Chronic Hepatitis B Treated With TDF
Brief Title: LDT Combined With TDF to Improve EGFR Decreasing in Patients With Chronic Hepatitis B Treated With TDF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chaoshuang Lin, Professor Lin, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 0000000
Record Dates: First submitted 2020-10-20; First posted 2020-11-25 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LDT Combined with TDF for Treatment: The patients take one tablet of LDTand one tablet of TDF every night and continue to 12 months.
- Only TAF treatment.: The patients take one tablet of TAF every night and continue to 12 months.

SUMMARY:
Chronic hepatitis B (CHB) is an important public health problem in the world. There are still more than 250 million chronic hepatitis B virus (CHB) infected people in the world. Its preventive effect has reached a relatively ideal effect, but its therapeutic effect still has great room for improvement.

Tenofovir(TDF) is the first-line antiviral treatment with good clinical efficacy. However, some patients who take TDF for a long time have different degrees of renal dysfunction, which limits the use of TDF in these patients.

Tenofovir Alafenamide Fumarate (TAF) has better plasma stability and stronger liver targeting, and reduces the side effects of renal function damage and bone mineral density reduction. Telbivudine (LDT), a nucleoside analogue, has the advantages of rapidly reducing HBV viral load and high HBeAg seroconversion rate.

In addition, prospective studies have shown that LDT can improve the estimated glomerular filtration rate (EGFR).Therefore, this study aims to explore the clinical study of LDT combined with TDF and TAF in patients treated with tenofovir and EGFR < 90ml / min / 1.72m².

DETAILED DESCRIPTION:
This is a multi-center, open-label clinical study. This study was aimed to explore the LDT combined with TDF and TAF in patients treated with TDF and EGFR < 90ml / min / 1.72m².The primary objectives of this study is as follows: To access the effectiveness and safety of 12-month treatment with LDT combined with TDF and only TAF in patients with CHC and cirrhosis in real-world clinical practice in Southern area of China. The proportion of participants with HBV DNA (DNA:Hepatitis B virus deoxyribonucleic acid)was evaluated. This study aims to enroll 200 patients with CHB in each treatment group. Patients with CHB having received the TAF previously but EGFR < 90ml / min / 1.72m² subsequently fulfills the indication of antiviral therapy will be administered with LDT combined with TDF and only TAF treatment. After 12-month treatment, all the patients will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. After TDF treatment, patients with eGFR<90ml/min/1.72m² and without obvious renal damage before taking the medicine switch to LDT combined with TDF, or switch to TAF treatment;
2. Patients had no obvious heart, lung and other important organ diseases in the past;
3. Patients have sign the informed consent form and complied with the study medication and follow-up plan.

Exclusion Criteria:

1. Co-infectious with hepatitis A, hepatitis C, hepatitis D, hepatitis E or HIV;
2. In the decompensated stage of liver cirrhosis, such as ascites, varicose bleeding or hepatic encephalopathy;
3. With malignant tumors (including hepatocellular carcinoma);
4. Concomitant with other liver diseases, such as alcoholic liver disease, autoimmune disease, or other systemic diseases involving the liver, such as hemochromatosis, Alpha-1 antitrypsin deficiency, or Wilson disease;
5. During the study period, chronic systemic steroid drugs are required or may be used under any medical conditions;
6. There are any other factors that the researcher thinks are not suitable for inclusion in the study, or that may affect the patient's participation or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mainly patients with decreased glomerular filtration rate after taking TDF and meeting the above inclusion criteria and not meeting any of the appeal exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
HBV DNA | 6 and 12 months
  Hepatitis B virus DNA is double-deoxyribonucleotide, which is a marker of hepatitis B virus replication.

SECONDARY OUTCOMES:
HBeAg seroconversion rate | 3,6,9,and 12 months
  HBeAg seroconversion rate means that HBeAg cannot be detected in the patient's serum but HBeAb can be detected.
Estimated glomerular filtration rate | 3,6,9,and 12 months
  Estimating the glomerular filtration rate can roughly reflect the condition of kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Chaoshuang Lin, Professor, Principal Investigator — Third Sun Yat Sen
Locations (1):
- Ermei Li, Guangzhou, Guangdong, China